CLINICAL TRIAL: NCT01717469
Title: Randomized Clinical Study to Assess the Safety and the Effects of Isolated Left Ventricular Pacing in Patients With Bradyarrhythmias
Brief Title: Safety and the Effects of Isolated Left Ventricular Pacing in Patients With Bradyarrhythmias
Acronym: SAFE-LVPACE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Duke University (Other)
Responsible Party: Principal Investigator, Roberto Costa, Associated Professor of Cardiovascular Surgery, MD PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE 00610412.2.0000.0068
Record Dates: First submitted 2012-09-30; First posted 2012-10-30 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Bradyarrhythmias; Arrhythmias; Atrioventricular Block; Ventricular Dysfunction; Cardiovascular Disease
Keywords: Pacemaker; Pacemaker implantation; Coronary sinus; Ventricular dysfunction; Right ventricular pacing; Left ventricular pacing
MeSH Terms: conditions — Bradycardia; Arrhythmias, Cardiac; Atrioventricular Block; Ventricular Dysfunction; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RV Pacing (Active Comparator): Right ventricular pacing
  Interventions: Device: Right ventricular pacing (Medtronic)
- LV Pacing (Experimental): Left ventricular pacing through coronary sinus tributaries
  Interventions: Device: Left ventricular pacing through coronary sinus tributaries (Attain StarFix)

INTERVENTIONS:
Device: Left ventricular pacing through coronary sinus tributaries (Attain StarFix) — Left ventricular pacing in patients with bradycardia
  Other Names: Attain StarFix® Model 4195 OTW Lead
  Arms: LV Pacing
Device: Right ventricular pacing (Medtronic) — Conventional right ventricular pacing in patients with bradycardia.
  Other Names: Right ventricular lead Medtronic 5076-58
  Arms: RV Pacing

SUMMARY:
Previous experimental and clinical studies have consistently suggested that right ventricular (RV) apical pacing has important adverse effects. Ventricular pacing, however, is required, and cannot be reduced in many patients with atrioventricular block. The SAFE-LVPACE study is a randomized controlled trial that compare the effects of conventional right ventricular (RV) pacing vs. left ventricular (LV) in patients with AV block.

DETAILED DESCRIPTION:
Over the past several years, there has been growing concern over the significant deleterious effects of RV pacing, including electromechanical dyssynchrony, proarrhythmia and development of heart failure (HF). However, it remains unclear whether pacing-related ventricular dyssynchrony can translate into significant LV structural changes and produce important clinical impairment in an average pacemaker population with compromised AV conduction. Alternatively, left ventricular pacing has been shown to minimize ventricular dyssynchrony and to improve symptoms and prognosis in patients with mild to moderated systolic HF and prolonged QRS duration.

This randomized controlled study is been conducted to compare the effects of conventional right ventricular (RV) pacing vs. left ventricular (LV) in patients with AV block. The hypothesis is that isolated LV pacing through the coronary sinus can be used safely and provide greater hemodynamic benefits to patients with AV block and normal ventricular function who require only the correction of heart rate.

Specifically, the investigator aims are to evaluate the safety, efficacy and the effects of left ventricular pacing using active-fixation coronary sinus lead-the Attain StarFix® Model 4195 OTW Lead, compared to right ventricular pacing in patients with implantation criteria for conventional pacemaker stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Pacemaker initial implant by transvenous approach
* Presence of AV block
* Presence of atrial fibrillation / atrial flutter with slow ventricular response
* Left ventricular systolic function > 0.40
* Subject agreed to participate and signed the consent form

Exclusion Criteria:

* Absence of venous access
* Impediment of venous access due to presence of intracardiac defects
* Impediment of venous access due to presence of tricuspid valve prosthesis
* Need for radiotherapy in the chest
* Presence of chest deformity
* Pregnancy
* Life expectancy of less than one year
* Contraindication to administration of iodinated contrast (creatinine > 3.0) Unable to attend the follow-up appointments

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2012-06; Primary Completion 2015-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Surgical success | Participants will be evaluated during the perioperative period and during the hospital stay, an expected average of 2 days
  Surgical success: absence of complications

SECONDARY OUTCOMES:
Echocardiographic and Clinical composite | Participants will be evaluated at 6 and 24 months after PM implantation
  Echocardiographic: ventricular dysfunction Clinical composite: all mortality, cardiovascular mortality, hospitalization, heart failure

OTHER OUTCOMES:
Quality of Life | Participants will be evaluated at 6 and 24 months after PM implantation
  Quality of life: improvement on quality of life scores measured by three questionnaires: 36-Item Short Form Health Survey (SF-36), a disease specific questionnaire for pacemaker patients (Aquarel) and Minnesota Living With Heart Failure (MLWHF).

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Costa, MD PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Heart Institute (InCor) do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil